CLINICAL TRIAL: NCT01788033
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2 Study of the Effects of XOMA 052 on Insulin Production in Subjects With Well-controlled Type 1 Diabetes
Brief Title: Effects of XOMA 052 on Insulin Production in Type 1 Diabetes
Acronym: LATE STAGE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: XOMA (US) LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EK-189/10
Record Dates: First submitted 2013-02-01; First posted 2013-02-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Diabetes Mellitus Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — gevokizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- XOMA 052 (Active Comparator): 0.3 mg/kg XOMA 052. Beginning on Day 0, each subject will receive one subcutaneous (SC) injection of study drug every 4 weeks for 12 weeks, a total of four injections
  Interventions: Drug: XOMA 052
- Placebo (Placebo Comparator): 0.3 mg/kg placebo. Beginning on Day 0, each subject will receive one subcutaneous (SC) injection of study drug every 4 weeks for 12 weeks, a total of four injections
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XOMA 052 — 0.3 mg/kg XOMA 052. Beginning on Day 0, each subject will receive one subcutaneous (SC) injection of study drug every 4 weeks for 12 weeks, a total of four injections
  Arms: XOMA 052
Drug: Placebo — 0.3 mg/kg Placebo. Beginning on Day 0, each subject will receive one subcutaneous (SC) injection of study drug every 4 weeks for 12 weeks, a total of four injections
  Arms: Placebo

SUMMARY:
To assess the effects of treatment with XOMA 052 on beta-cell function and insulin production in subjects with well-controlled Type 1 diabetes. The safety, tolerability, and pharmacokinetics (PK) of XOMA 052 will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes (American Diabetes Association [ADA] criteria) of > 2 year duration that is judged to be stable by the investigator
* No clinically significant change in treatment regimen for T1D (defined as a 20% change) during the 3 months prior to Screening
* Age ≥ 18 years and ≤ 55 years
* HbA1c < 7.5% for the previous two measurements including the measurement taken at Screening (both measurements must occur within 6 months prior to enrollment)
* Positive glutamate decarboxylase-65 (GAD65) and/or IA-2 auto-antibodies
* Body-mass index (BMI) > 18 and < 28 kg/m2
* Willingness to maintain current doses/regimens of vitamins and dietary supplements through the end of the study
* For subjects with reproductive potential, a willingness to use contraceptive measures adequate to prevent the subject or the subject's partner from becoming pregnant during the study. Adequate contraceptive measures include hormonal methods used for two or more cycles prior to Screening (e.g., oral contraceptive pills, contraceptive patch, or contraceptive vaginal ring), double barrier methods (e.g., contraceptive sponge, diaphragm used in conjunction with contraceptive foam or jelly, and condom used in conjunction with contraceptive foam or jelly), intrauterine methods (IUD), sterilization (e.g., tubal ligation or a monogamous relationship with a vasectomized partner), and abstinence.
* For females receiving hormone replacement therapy (including but not limited to oral contraceptives), must have been on a stable regimen for ≥ 6 months prior to Screening. Hormone therapy must not be initiated during the study

Exclusion Criteria:

* Signs of current infection or history of infection during the 3 months prior to Day 0
* Known to be positive for Hep B surface antigen (HBsAg), Hep C virus (HCV), or HIV
* History of tuberculosis (TB) or positive PPD test. A subject who has had a positive PPD test but has completed a course of treatment for tuberculosis, had a documented vaccination against tuberculosis, or had a negative QuantiFERON®-TB test result is eligible.
* High sensitivity C-reactive protein (hs-CRP) > 10 mg/L
* Presence of foot, leg, or decubitus ulcers
* Neutropenia
* Anemia
* Clinically significant kidney or liver disease
* From 1 week prior to Screening, use of anti-inflammatory therapy other than aspirin ≤ 100 mg/day or up to 5 consecutive days of treatment with non-steroidal anti-inflammatory drugs (NSAIDs) for treatment of an acute illness
* Current immunosuppressive treatment or documented immunodeficiency
* History of severe allergic or anaphylactic reactions
* History of asthma requiring systemic corticosteroid therapy
* Coronary intervention or hospitalization for cardiovascular condition within 12 months prior to Day 0
* Uncontrolled hypertension
* History of congestive heart failure
* History of a coronary event within 12 months prior to Screening
* Female subjects who are pregnant, planning to become pregnant during the course of the study, have recently delivered (within 3 month of Screening), or are breast-feeding
* History of malignancy within 5 years prior to study entry other than carcinoma in situ of the cervix or thyroid, or adequately treated, non-metastatic squamous or basal cell carcinoma of the skin
* Receipt of a live (attenuated) vaccine within 3 months prior to Screening
* Use of any other investigational drug within 30 days prior to enrollment or within 5 half-lives of the investigational drug, whichever is longer
* Any condition which, in the opinion of the investigator, would jeopardize the subject's safety following exposure to the study drug
* Any condition (e.g., psychiatric illness) or situation that may compromise the ability of the subject to give written informed consent, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2009-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
C-peptide level | incremental AUC over 120 minutes during the MMTT at Day 112 compared to baseline (Day 0 pre-dose

SECONDARY OUTCOMES:
Change in insulin requirements | 3-day average daily insulin dose at baseline (Day -3 through Day -1) compared to Day 112 (Day 109 through Day 111)
HbA1c levels | from baseline (Day 0 pre-dose) at Day 112
fasting glucose | from baseline (Day 0 pre-dose) at Day 112
fasting glucagon | from baseline (Day 0 pre-dose) at Day 112
cortisol | from baseline (Day 0 pre-dose) at Day 112
markers of systemic inflammation (Interleukin-6, Interleukin-8, Tumor Necrosis Factor α, hs-CRP) | from baseline (Day 0 pre-dose) at Day 112
adipokines | from baseline (Day 0 pre-dose) at Day 112
meal-stimulated Glucagon like peptide-1 | AUC over 120 minutes at Day 112 compared to baseline (Day 0 pre-dose)
meal-stimulated gastric inhibitory polypeptide | AUC over 120 minutes at Day 112 compared to baseline (Day 0 pre-dose)
lipids profile | from baseline (Day 0 pre-dose) at Day 112
Change in fatigue according to the Fatigue Scale for Motor and Cognitive Functions (FSMC) questionnaire | from baseline at Day 112
Anti XOMA 052 Antibodies | from baseline (Day 0 pre-dose) at Day 112
Number of Adverse Events | from baseline (Day 0 pre-dose) at Day 364

CONTACTS AND LOCATIONS:
Overall Officials: Marc Donath, Prof., Study Chair — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Basel, Switzerland